CLINICAL TRIAL: NCT04981249
Title: Risk of Severe COVID-19, Taking Into Account Multimorbidity Patterns, as Well as Other Clinical and Sociodemographic Variables. Big Data Mrisk-COVID Project
Brief Title: Chronic Multimorbidity Patterns in Relation to COVID-19 Severe Infection
Acronym: Mrisk-COVID
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Agència de Qualitat i Avaluació Sanitàries (Other Government); Instituto Aragones de Ciencias de la Salud (Other Government)
Responsible Party: Principal Investigator, Marisa Baré, MD, MPH, PhD, Coordinator, Corporacion Parc Tauli
Other Study IDs: CIR 2020/023
Record Dates: First submitted 2021-07-27; First posted 2021-07-28 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Covid-19; Chronic Disease
Keywords: Multimorbidity; Cluster analysis; Covid-19
MeSH Terms: conditions — COVID-19; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to analyze the patterns of chronic multimorbidity of a cohort of Covid-19 patients, and to assess the relation between the patterns and the development of severe infection or mortality.

DETAILED DESCRIPTION:
This is a Big Data study that aims to establish the multimorbidity (MM) clusters of a cohort of Covid-19 patients, and assess their potential relation with severe infection or mortality. Databases of demographic information and complete medical records from the cohort will be provided by the Agency for Health Quality and Assessment of Catalonia (AQuAS). Data will be collected and integrated in a complete database in order to define the study variables: multimorbidity patterns, COVID-19 severe infection and COVID-19 associated mortality. The population will be stratified by sex and age (21-45, 46-65, 66-80 and 81-95 years). Diagnoses from primary care and hospitals will be filtered and classified using the Chronic Condition Indicator v.2021 and the Clinical Classification Software v.2021 [1], in order to identify the Chronic Conditions (CC) of the patients. CC with prevalence >2% in each age-sex strata will be subjected to a fuzzy c-means clustering analysis. The final number of clusters in each age-sex group will be determined under the clinical criteria of the research group members. Percentages of patients that suffered severe Covid-19 infection or death in each cluster will be calculated. Bivariate statistical analysis comparing the demographic data and the cluster distribution with severe infection and mortality will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Positive results of Covid-19 laboratory tests
* Covid-19 related clinical profile verified by healthcare professionals

Exclusion Criteria:

* Male >90 years
* Females >95 years

Ages: 21 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Confirmed or suspected Covid-19 patients from the first wave of the pandemic, aged >20 years, residing in a healthcare region of about 400.000 inhabitants in a Northeast region of Spain (Vallès Occidental Est, Catalonia, Spain).
Sampling Method: Non-Probability Sample
Enrollment: 14286 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Covid-19 severe infection | From 27-February-2020 to 15-June-2020
  Severe COVID-19 infection was defined as the occurrence of at least one of the following conditions during any of the registered COVID-19 episodes: severe respiratory affection (including insufficiency, failure, or distress); use of respiratory support (including mechanical ventilation or oxygen therapy); septic shock; multiple organ failure (the combination of respiratory failure and any other organ failure); inflammatory response; admission to intensive care unit; and mortality.
Covid-19 mortality | From 27-February-2020 to 15-June-2020
  Death associated to COVID-19 infection episode

CONTACTS AND LOCATIONS:
Locations (1):
- Corporacio Parc Taulí, Sabadell, Spain

REFERENCES:
- [Derived] Lleal M, Corral-Vazquez C, Bare M, Comet R, Herranz S, Baigorri F, Gimeno-Miguel A, Raurich M, Fortia C, Navarro M, Poblador-Plou B, Bare M. Multimorbidity patterns in COVID-19 patients and their relationship with infection severity: MRisk-COVID study. PLoS One. 2023 Aug 31;18(8):e0290969. doi: 10.1371/journal.pone.0290969. eCollection 2023. PMID 37651465
- See also: Agency for Healthcare Research and Quality. Rockville. MD. Healthcare Cost and Utilization Project (HCUP) — https://www.hcup-us.ahrq.gov/home.jsp